CLINICAL TRIAL: NCT05179408
Title: Telerehabilitation for Veteran Lung Cancer Survivors Following Curative Intent Therapy
Brief Title: Targeted Telerehabilitation Following Curative Intent Therapy of Lung Cancer
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: F3661-W; RX003661 (Other Grant/Funding Number: Department of Veterans Affairs)
Record Dates: First submitted 2021-12-16; First posted 2022-01-05 (Actual); Last update posted 2026-01-27 (Actual); Status verified 2026-01

CONDITIONS: Lung Cancer; Cancer Survivors
Keywords: Rehabilitation; Exercise training; Mindfulness training; Survivorship; US Veterans; Telemedicine
MeSH Terms: conditions — Lung Neoplasms | interventions — Waiting Lists

STUDY DESIGN:
Intervention Model Description: This project will evaluate multi-targeted telerehabilitation with Veteran lung cancer survivors following curative intent therapy. Targets include: 1) inspiratory muscle training + walking promotion to reduce dyspnea and improve physical activity; 2) resistance training to reduce cancer-related fatigue and improve social/role functioning; and 3) mindfulness training to reduce fear of cancer recurrence and cancer-related anxiety.
Who Masked: Outcomes Assessor
Masking Description: The outcome assessor will be blinded to participant allocation group.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Targeted telerehabilitation (Experimental): Participant-chosen targets: 1) inspiratory muscle training + walking (to reduce dyspnea and improve physical activity/endurance; 2) resistance training (to reduce fatigue and improve role/social function; 3) mindfulness training (to reduce fear of cancer recurrence and anxiety)
  Interventions: Behavioral: Targeted-telerehabilitation
- Waitlist (Active Comparator): 8-week waiting period prior to participating in targeted telerehabilitation
  Interventions: Behavioral: Waitlist

INTERVENTIONS:
Behavioral: Targeted-telerehabilitation — Participant-chosen targets: 1) inspiratory muscle training + walking (to reduce dyspnea and improve physical activity/stept count; 2) resistance training (to reduce fatigue and improve role/social function; 3) mindfulness training (to reduce fear of cancer recurrence and anxiety)
  Arms: Targeted telerehabilitation
Behavioral: Waitlist — 8-week waiting period prior to targeted telerehabilitation
  Arms: Waitlist

SUMMARY:
Lung cancer is the second-most commonly diagnosed cancer among U.S. Veterans. Substantial advances have been made in early detection through screening and treatment. The longevity of Veterans following lung cancer diagnosis and treatment has increased. Following treatment however, many Veterans experience increased symptom burden, particularly in shortness of breath, fatigue, and fear/anxiety about lung cancer, and impairments in physical and psychosocial functioning. Rehabilitation services are needed to address these survivorship challenges. This study will evaluate multi-targeted telerehabilitation with Veterans following lung cancer treatment, with goals to reduce symptom burden, improve physical and psychosocial function, and enhance health-related quality of life. This research will also develop the career of a physician researcher to acquire expertise in rehabilitation for many Veteran survivors of lung and other cancers.

DETAILED DESCRIPTION:
Lung cancer is the second-most commonly diagnosed cancer among U.S. Veterans - over 8,200 incident cases are diagnosed each year. Approximately 50% of lung cancers are diagnosed at stage I-III and therefore eligible for curative intent therapy. Survival rates among Veterans with early stage lung cancer have increased along with advances in surgical and radiation techniques. Following curative intent therapy, many Veterans experience physical function loss and increased symptom burden, particularly in dyspnea, fatigue, and fear/anxiety. Approaches are needed to improve their physical and psychosocial function and health-related quality of life (HRQL). We hypothesize that multi-targeted telerehabilitation could mitigate these HRQL impairments. Therefore, we will conduct a pilot randomized trial to examine the (a) feasibility, (b) acceptability, (c) safety, and (d) explore the effects of multi-targeted telerehabilitation with these patients. Participants (N=30-40) will be randomized (3:1) to receive 8 weeks of participant-chosen targeted telerehabilitation (experimental arm) or waitlist condition (control arm). Feasibility will be assessed by enrollment, adherence, retention and exploratory effects by linear mixed effects models comparing changes in patient-centered outcomes from baseline to end-of-intervention between groups: dyspnea, daily step count, fatigue, role/social function, fear/anxiety, and HRQL. This project will provide pilot data and training for an early career physician investigator to establish independence, with a goal of a large-scale, preference-informed randomized trial of targeted and patient-centered telerehabilitation, to improve the physical and psychosocial function, independence, and HRQL of Veteran lung cancer survivors following curative intent therapy.

ELIGIBILITY:
Inclusion Criteria:

* Adult Veterans with a history of stage I-III A/B lung cancer, and
* Completed curative intent therapy (i.e., lung cancer resection surgery, definitive radiation, or concurrent chemoradiation) within 1-6 months

Exclusion Criteria:

* Adult Veterans with any comorbid conditions that preclude participation in exercise and telerehabilitation:
* Orthopedic conditions (e.g., bilateral below-knee amputation), or
* Severe cardiopulmonary disease (e.g., unstable arrhythmias including ventricular tachycardia, heart failure with systolic ejection fraction < 25%, chronic hypoxemia needing > 5 L/min oxygen supplementation at rest), or
* Inability to follow directions or provide informed consent (e.g., moderate to severe dementia), or
* Enrolled in hospice, or
* With an estimated life expectancy of < 6 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2026-01-12 (Actual); Primary Completion 2027-03-30 (Estimated); Study Completion 2027-03-30 (Estimated)

PRIMARY OUTCOMES:
Health-related quality of life (HRQL) | Difference in changes in HRQL between baseline and end-of-intervention (8 weeks)
  Global health-related quality of life (EORTC QLQ C30 global/QoL subscale)

SECONDARY OUTCOMES:
Dysnea and physical activity (participant-chosen) | Differences in changes in UCSD SOBQ and average steps/day between baseline and end-of-intervention (8 weeks)
  University of California Shortness of Breath Questionnaire (UCSD SOBQ) and Fitbit stepcount
Cancer-related function (participant chosen) | Difference in changes in PROMIS-SF Cancer Function 3D Profile between baseline and end-of-intervention (8 weeks)
  PROMIS-SF Cancer Function 3D Profile (fatigue, role, and social function)
Fear of Cancer Recurrence and Cancer-related Anxiety (participant chosen) | Difference in changes in FCR and PROMIS-SF Anxiety 8a between baseline and end-of-intervention (8 weeks)
  Fear of Cancer Recurrence (FCR) and PROMIS-SF Anxiety 8a

CONTACTS AND LOCATIONS:
Overall Officials: Duc M. Ha, MD MAS, Principal Investigator — Rocky Mountain Regional VA Medical Center, Aurora, CO
Locations (1):
- Rocky Mountain Regional VA Medical Center, Aurora, CO, Aurora, Colorado, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ha D, Ries AL, Lippman SM, Fuster MM. Effects of curative-intent lung cancer therapy on functional exercise capacity and patient-reported outcomes. Support Care Cancer. 2020 Oct;28(10):4707-4720. doi: 10.1007/s00520-020-05294-3. Epub 2020 Jan 21. PMID 31965306
- [Background] Ha D, Ries AL, Mazzone PJ, Lippman SM, Fuster MM. Exercise capacity and cancer-specific quality of life following curative intent treatment of stage I-IIIA lung cancer. Support Care Cancer. 2018 Jul;26(7):2459-2469. doi: 10.1007/s00520-018-4078-4. Epub 2018 Feb 10. PMID 29429006
- [Background] Ha D, Kerr J, Ries AL, Fuster MM, Lippman SM, Murphy JD. A Model-Based Cost-Effectiveness Analysis of an Exercise Program for Lung Cancer Survivors After Curative-Intent Treatment. Am J Phys Med Rehabil. 2020 Mar;99(3):233-240. doi: 10.1097/PHM.0000000000001281. PMID 31361623
- [Background] Ha DM, Zeng C, Chan ED, Gray M, Mazzone PJ, Samet JM, Steiner JF. Association of Exercise Behavior with Overall Survival in Stage I-IIIA Lung Cancer. Ann Am Thorac Soc. 2021 Jun;18(6):1034-1042. doi: 10.1513/AnnalsATS.202003-235OC. PMID 33326358
- [Background] Ha DM, Prochazka AV, Bekelman DB, Stevens-Lapsley JE, Studts JL, Keith RL. Modifiable factors associated with health-related quality of life among lung cancer survivors following curative intent therapy. Lung Cancer. 2022 Jan;163:42-50. doi: 10.1016/j.lungcan.2021.11.012. Epub 2021 Dec 2. PMID 34896804
- [Background] Ha DM, Comer A, Dollar B, Bedoy R, Ford M, Gozansky WS, Zeng C, Arch JJ, Leach HJ, Malhotra A, Prochazka AV, Keith RL, Boxer RS. Telemedicine-based inspiratory muscle training and walking promotion with lung cancer survivors following curative intent therapy: a parallel-group pilot randomized trial. Support Care Cancer. 2023 Sep 1;31(9):546. doi: 10.1007/s00520-023-07999-7. PMID 37656252
- [Background] Ha DM, Nunnery MA, Klocko RP, Haverhals LM, Bekelman DB, New ML, Randhawa SK, Stevens-Lapsley JE, Studts JL, Prochazka AV, Keith RL. Lung cancer survivors' views on telerehabilitation following curative intent therapy: a formative qualitative study. BMJ Open. 2023 Jun 23;13(6):e073251. doi: 10.1136/bmjopen-2023-073251. PMID 37355268
- [Background] Ha DM, Prochazka AV, Bekelman DB, Stevens-Lapsley JE, Chan ED, Keith RL. Association of Leisure-Time Physical Activity With Health-Related Quality of Life Among US Lung Cancer Survivors. JNCI Cancer Spectr. 2021 Jan 23;5(1):pkaa118. doi: 10.1093/jncics/pkaa118. eCollection 2021 Feb. PMID 35075444
- [Background] Ha D, Ries AL. Characterization of Dyspnea in Veteran Lung Cancer Survivors Following Curative-Intent Therapy. J Cardiopulm Rehabil Prev. 2020 Mar;40(2):120-127. doi: 10.1097/HCR.0000000000000464. PMID 31592931
- [Background] Ha D, Malhotra A, Ries AL, O'Neal WT, Fuster MM. Heart rate variability and heart rate recovery in lung cancer survivors eligible for long-term cure. Respir Physiol Neurobiol. 2019 Nov;269:103264. doi: 10.1016/j.resp.2019.103264. Epub 2019 Jul 31. PMID 31376471
- [Background] Bade BC, Faiz SA, Ha DM, Tan M, Barton-Burke M, Cheville AL, Escalante CP, Gozal D, Granger CL, Presley CJ, Smith SM, Chamberlaine DM, Long JM, Malone DJ, Pirl WF, Robinson HL, Yasufuku K, Rivera MP. Cancer-related Fatigue in Lung Cancer: A Research Agenda: An Official American Thoracic Society Research Statement. Am J Respir Crit Care Med. 2023 Mar 1;207(5):e6-e28. doi: 10.1164/rccm.202210-1963ST. PMID 36856560
- [Background] Parshall MB, Schwartzstein RM, Adams L, Banzett RB, Manning HL, Bourbeau J, Calverley PM, Gift AG, Harver A, Lareau SC, Mahler DA, Meek PM, O'Donnell DE; American Thoracic Society Committee on Dyspnea. An official American Thoracic Society statement: update on the mechanisms, assessment, and management of dyspnea. Am J Respir Crit Care Med. 2012 Feb 15;185(4):435-52. doi: 10.1164/rccm.201111-2042ST. PMID 22336677
- [Background] Rochester CL, Alison JA, Carlin B, Jenkins AR, Cox NS, Bauldoff G, Bhatt SP, Bourbeau J, Burtin C, Camp PG, Cascino TM, Dorney Koppel GA, Garvey C, Goldstein R, Harris D, Houchen-Wolloff L, Limberg T, Lindenauer PK, Moy ML, Ryerson CJ, Singh SJ, Steiner M, Tappan RS, Yohannes AM, Holland AE. Pulmonary Rehabilitation for Adults with Chronic Respiratory Disease: An Official American Thoracic Society Clinical Practice Guideline. Am J Respir Crit Care Med. 2023 Aug 15;208(4):e7-e26. doi: 10.1164/rccm.202306-1066ST. PMID 37581410
- [Background] Shaw J, Kamphuis H, Sharpe L, Lebel S, Smith AB, Hulbert-Williams N, Dhillon HM, Butow P. Setting an International Research Agenda for Fear of Cancer Recurrence: An Online Delphi Consensus Study. Front Psychol. 2021 Feb 22;12:596682. doi: 10.3389/fpsyg.2021.596682. eCollection 2021. PMID 33692719